CLINICAL TRIAL: NCT00183313
Title: Improving Primary Care in Patients With Mental Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Benjamin Druss, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00002164; R01MH070437 (NIH); DSIR 82-SEPC
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Mental Disorders
Keywords: Mental Health; Primary health care; Case management
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive nurse case management intervention
  Interventions: Behavioral: Nurse case management
- 2 (Active Comparator): Participants will receive usual care
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Nurse case management — Nurse case management is a population-based medical case management program to improve the delivery of primary medical care to patients with serious mental illness in a Community Mental Health Center (CMHC) in Atlanta GA. The treatment draws on elements from the primary care, nursing case management, chronic disease, health behavior change literature, and from the study team's experience in integrating primary care services for patients with serious mental illnesses.
  Arms: 1
Behavioral: Usual care — Usual care includes standard mental health services.
  Arms: 2

SUMMARY:
This study will determine the effectiveness of medical case management in improving the medical care of people with mental disorders or substance abuse problems.

DETAILED DESCRIPTION:
Poor quality of care may contribute to impaired health status and increased mortality in individuals with serious mental disorders and substance abuse problems; interventions designed to improve medical care for this population need to be developed. This study will develop a population-based medical case management model for improving the primary medical care of patients at an inner city community mental health center.

This study will last 2 years. Participants will be randomly assigned to receive medical case management or standard of care (typically drug and behavioral therapy) for 2 years. Participants in the case management group will receive help in overcoming barriers to receiving primary care. Participants will also undergo 5 interviews over the 2-year study duration, and have annual chart reviews. Results of the interviews will be used to assess quality of primary care, service use, health outcomes, psychiatric symptoms, and substance use.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mental illness or substance abuse
* Patient at Florida Hall (Grady Health Systems)

Exclusion Criteria:

* Current use of medical case management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2004-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Quality of primary medical care | Measured over 2 years

SECONDARY OUTCOMES:
Health status | Measured over 2 years
Psychiatric symptoms | 2004-2009
Costs | 2004-2009

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin G. Druss, MD, MPH, Principal Investigator — Emory University; Silke A. von Esenwein, MA, Study Director — Emory University
Locations (2):
- United States (2):
  - Grady Health Systems, Atlanta, Georgia
  - Emory University, Atlanta, Georgia

REFERENCES:
- [Derived] Druss BG, von Esenwein SA, Compton MT, Rask KJ, Zhao L, Parker RM. A randomized trial of medical care management for community mental health settings: the Primary Care Access, Referral, and Evaluation (PCARE) study. Am J Psychiatry. 2010 Feb;167(2):151-9. doi: 10.1176/appi.ajp.2009.09050691. Epub 2009 Dec 15. PMID 20008945